CLINICAL TRIAL: NCT03436069
Title: Identification de Nouveaux Marqueurs Pronostiques Des Cancers du Sein
Brief Title: Identification of New Prognostic Markers for Breast Cancer.
Acronym: PROBREAST
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC17.172; 2017-A01740-53 (Other: ID RCB)
Record Dates: First submitted 2017-12-14; First posted 2018-02-19 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Breast Cancer
Keywords: Breast cancer; biomarkers; prognostic; ectopic gene expression; expression profile; tissue-specific genes; response to treatment
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — The research uses blood samples and biopsies made at diagnosis or during surgical resection of the tumor for gene or protein expression analysis (RNA and protein extraction).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Conventional treatment protocols of breast cancer

SUMMARY:
Candidate markers have been identified thanks to an original approach developed by our research team aiming at detecting ectopic gene expression using public pan-genomic breast cancer data. The same approach had already been used and validated in lung tumors, leukemias and lymphomas. The main objective of the present research is to use tumor samples from patients in a retrospective and prospective cohort to test and validate the relevance of these prognostic markers in breast cancer.

DETAILED DESCRIPTION:
Following a diagnosis of breast cancer, the most immediate challenges in patient management are the determination of prognosis and the identification of the most appropriate neoadjuvant and adjuvant systemic therapy. Indicators to assess the risk of relapse or metastasis during treatment are still largely insufficient, a situation which does not allow to precisely adjust the treatment, often leading to heavy side effects. In order to minimize the side effects and risks of therapies, it is therefore necessary to discover new markers which would enable us to reliably assess the prognosis of patients diagnosed with breast cancer.

The approach used here for discovering new prognostic markers is based on an original strategy developed by the researchers associated with this project and published in the respective contexts of lung cancer, acute lymphoblastic leukemia and lymphoma. Indeed, genetic abnormalities and deregulation of the systems controlling the expression of specific gene programs not only lead to the abnormal extinction of normally active genes, but is also responsible for the aberrant activation of genes that normally should remain silent. The investigators have recently demonstrated that any type of malignancy is associated with the ectopic expression of these normally silent genes, including genes of the male germline. The in-depth study of these aberrant gene expressions and the search for correlations and associations with the clinical and biological data of the tumors show that the expression of some of these genes and the presence of their products are good indicators of tumor aggressiveness.

The investigators propose here to apply the same approach for the search for new prognostic markers in the case of breast cancer. A prior analysis of breast tumors, of which transcriptome data are publicly available, has identified a number of tissue-specific genes, including the germline and placenta genes, frequently activated in breast cancer. Based on our past observations, our hypothesis is that some of them may directly reflect the level of tumor aggressiveness and could therefore be used as prognostic biomarkers.

The objective of this work will be to look for the prognostic value of these genes by using the samples collected in this cohort of patients to detect their activation and to correlate these aberrant activations with the anatomopathological data of the tumor, as well as to the clinico-biological data and patient follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Adult female patients with breast cancer

Exclusion Criteria:

* Presence of another cancer, excluding basal cell cancers or pre-neoplastic lesions of the cervix.
* Subject under guardianship or subject deprived of liberty
* Impossibility of collecting information on exposure (subjects recently arrived in France, foreign language, etc.)
* Male patients

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult female patients with breast cancer
Sampling Method: Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2011-01 (Actual); Primary Completion 2033-12-31 (Estimated); Study Completion 2033-12-31 (Estimated)

PRIMARY OUTCOMES:
Study of ectopic gene expression to define new prognostic biomarkers in breast cancer | 12 years, with evaluation every 3 years
  The overall survival and disease-free survival of patient with breast cancers will be analyzed in terms of gene expression change in order to identify new prognostic biomarkers.

SECONDARY OUTCOMES:
Study of response to neoadjuvant treatments of breast cancer assessed from anatomopathological data. | 12 years, with evaluation every 3 years
  Evaluation of a response rate after neoadjuvant chemotherapy according to RECIST criteria

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Cécile PHILIPPE, Dr, Principal Investigator — University Hospital, Grenoble; Mireille MOUSSEAU, Pr, Study Director — Grenoble Alpes University Hospital
Locations (1):
- Anne-Cécile PHILIPPE, Grenoble, France

REFERENCES:
- [Background] Wang J, Mi JQ, Debernardi A, Vitte AL, Emadali A, Meyer JA, Charmpi K, Ycart B, Callanan MB, Carroll WL, Khochbin S, Rousseaux S. A six gene expression signature defines aggressive subtypes and predicts outcome in childhood and adult acute lymphoblastic leukemia. Oncotarget. 2015 Jun 30;6(18):16527-42. doi: 10.18632/oncotarget.4113. PMID 26001296
- [Background] Le Bescont A, Vitte AL, Debernardi A, Curtet S, Buchou T, Vayr J, de Reynies A, Ito A, Guardiola P, Brambilla C, Yoshida M, Brambilla E, Rousseaux S, Khochbin S. Receptor-Independent Ectopic Activity of Prolactin Predicts Aggressive Lung Tumors and Indicates HDACi-Based Therapeutic Strategies. Antioxid Redox Signal. 2015 Jul 1;23(1):1-14. doi: 10.1089/ars.2013.5581. Epub 2014 Mar 6. PMID 24512221
- [Background] Emadali A, Rousseaux S, Bruder-Costa J, Rome C, Duley S, Hamaidia S, Betton P, Debernardi A, Leroux D, Bernay B, Kieffer-Jaquinod S, Combes F, Ferri E, McKenna CE, Petosa C, Bruley C, Garin J, Ferro M, Gressin R, Callanan MB, Khochbin S. Identification of a novel BET bromodomain inhibitor-sensitive, gene regulatory circuit that controls Rituximab response and tumour growth in aggressive lymphoid cancers. EMBO Mol Med. 2013 Aug;5(8):1180-95. doi: 10.1002/emmm.201202034. Epub 2013 Jul 4. PMID 23828858
- [Background] Rousseaux S, Debernardi A, Jacquiau B, Vitte AL, Vesin A, Nagy-Mignotte H, Moro-Sibilot D, Brichon PY, Lantuejoul S, Hainaut P, Laffaire J, de Reynies A, Beer DG, Timsit JF, Brambilla C, Brambilla E, Khochbin S. Ectopic activation of germline and placental genes identifies aggressive metastasis-prone lung cancers. Sci Transl Med. 2013 May 22;5(186):186ra66. doi: 10.1126/scitranslmed.3005723. PMID 23698379
- [Background] Reynoird N, Schwartz BE, Delvecchio M, Sadoul K, Meyers D, Mukherjee C, Caron C, Kimura H, Rousseaux S, Cole PA, Panne D, French CA, Khochbin S. Oncogenesis by sequestration of CBP/p300 in transcriptionally inactive hyperacetylated chromatin domains. EMBO J. 2010 Sep 1;29(17):2943-52. doi: 10.1038/emboj.2010.176. Epub 2010 Jul 30. PMID 20676058